CLINICAL TRIAL: NCT04371185
Title: A Randomized, Double-blinded, Single-dose, 3-arms Parallel, Comparative Study to Evaluate the Pharmacokinetics and Safety of BAT2206 Injection vs Ustekinumab Injection (Stelara) in Healthy Chinese Male Subjects
Brief Title: Comparative Study to Evaluate the Pharmacokinetics of BAT2206 vs Stelara® in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAT-2206-001-CR
Record Dates: First submitted 2020-03-23; First posted 2020-05-01 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BAT2206 injection (Experimental): 45mg; subcutaneous injection
  Interventions: Drug: BAT2206
- Stelara(US-licensed) (Active Comparator): 45mg; subcutaneous injection
  Interventions: Drug: Stelara(US-licensed)
- Stelara(EU-licensed) (Active Comparator): 45mg; subcutaneous injection
  Interventions: Drug: Stelara(EU-licensed)

INTERVENTIONS:
Drug: BAT2206 — 45mg/0.5 ml; single dose；prefilled syringe; subcutaneous injection
  Arms: BAT2206 injection
Drug: Stelara(US-licensed) — 45mg/0.5 ml; single dose；prefilled syringe; subcutaneous injection
  Other Names: Ustekinumab
  Arms: Stelara(US-licensed)
Drug: Stelara(EU-licensed) — 45mg/0.5 ml; single dose；prefilled syringe; subcutaneous injection
  Other Names: Ustekinumab
  Arms: Stelara(EU-licensed)

SUMMARY:
It is a randomized, double-blinded, single-dose, 3-arm parallel, comparative study to evaluate the pharmacokinetics, safety and immunogenicity of BAT2206 Injection vs Stelara® (EU-licensed and US-licensed) in healthy Chinese male subjects. A total of 270 healthy male subjects are planned to be included and randomized at a ratio of 1:1:1 to receive single 45mg/0.5ml BAT2206 Injection or Stelara® (EU-licensed and US-licensed).

DETAILED DESCRIPTION:
The study has a screening period of 14 days. PK blood samples will be collected from subjects to determine the serum concentration of Ustekinumab, thus to evaluate the similarity of the pharmacokinetics of the three study drugs.

The investigator will perform safety evaluation for vital signs, physical examinations, injection site reaction, ECG, clinical laboratory tests and adverse events throughout the study. Immunogenicity evaluation (ADA, ADA titration and nAb) will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Chinese male healthy subjects aged from 18 to 55 years (including the boundary value)；
* BMI between 18-28kg/m2 (including boundary value) and body weight between 55-85kg;
* Normal physical examination results or abnormal with no clinical significance according to the doctor's judgment;
* The subject (including partner) has no pregnancy plan or sperm donation plan during the whole trial period and within 6 months after the completion of the study, and voluntarily adopts effective contraceptive measures;
* Sign the informed consent before joining the study, and fully understand the content, process and possible risks;
* Willing and able to comply with the visits and treatments of the trial protocol.

Exclusion Criteria:

* Clinical laboratory examination results are abnormal and with clinical significance, or other clinical findings indicate diseases with clinical significance within one year prior to screening;
* ECG is abnormal and has clinical significance (judged by the investigator);
* With active infection within two months before screening, including acute and chronic infection and local infection;
* Hepatitis B and/or Hepatitis C; or HIV antigen/antibody positive; or Treponema pallidum antibody positive;
* Having taken any prescription drug, over-the-counter drug, any vitamin product or herbal medicine within 28 days before screening (or within 5 half-lives of the above drugs, whichever is longer);
* Having participated in drug clinical trials within 3 months before the study administration, or planning to participate in other drug clinical trials during the study period;
* Acute disease occurred or with concomitant medication from the screening to use of the study drug; major injury or surgery or fracture occurred within 4 weeks before enrollment, or surgery was planned during the study;
* Having used ustekinumab, anti-tumor necrosis factor (TNF) or interleukin (IL) targeting agents, or having used any biological products or monoclonal antibodies within 3 months before screening;
* Any immunoglobulin biologicals were used one year prior to screening;
* Having received within 12 weeks prior to initiating treatment or planning to receive live virus or live vaccines during the study;
* Suspected or confirmed as allergic constitution (allergic to variety of drugs or food), or allergic to ustekinumab, or severe allergic or allergic reaction to monoclonal antibody;
* Blood donation or massive blood loss (> 450 ml) within 3 months before using the study drug, or planning to donate blood during the study, or having received blood transfusion within 8 weeks before screening;
* Employees or relatives of all investigators, clinical centers, clinical research organizations or sponsors cannot be included in the group;
* Subjects considered unsuitable by the investigators.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 270 (Actual)
Dates: Start 2020-08-08 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics Endpoint: Peak plasma concentration (Cmax) | 0-4months
Pharmacokinetics Endpoint: Area under the plasma concentration versus time curve (AUC0-inf) | 0-4months

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, Principal Investigator — the First Hospital of Jinlin University
Locations (1):
- The First Hospital of Jilin University, Jilin, China

IPD SHARING:
Plan to Share IPD: No
Only one site study

REFERENCES:
- [Derived] Wu M, Li X, Yang D, Wang M, Zhang H, Li C, Mai J, Yang L, Qi Y, Yu JC, Yang X, Wang Z, Gu C, Ding Y. Comparison of Pharmacokinetic Similarity, Immunogenicity, and Safety of Ustekinumab and BAT2206 in Healthy Chinese Male Subjects in a Double-Blind, Randomized, Single-Dose, Parallel-Group Phase I Trial. BioDrugs. 2023 Jan;37(1):89-98. doi: 10.1007/s40259-022-00563-5. Epub 2022 Nov 22. PMID 36417156